CLINICAL TRIAL: NCT00527345
Title: Children's Exposure and Health Effects From Diesel Exhaust Before and After Switch of Schoool Bus Fleets
Brief Title: Children's Exposures/Health Effects/Diesel Exhaust
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 12657-CP-001; R01ES012657 (NIH)
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Asthma; Airway Inflammation
Keywords: Asthma; Diesel exhaust
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: children riding retrofitted school buses or private cars
- 2: children riding old buses who will change to retrofitted buses during the first or second year of the study
- 3: children who ride old diesel buses through the study

SUMMARY:
The contribution of diesel exhaust (DE) to health, especially children's health, is of tremendous public health interest. DE has been associated with worsening asthma and allergies, among other important health effects. Reducing DE exposures has become a major regulatory initiative, and federal, state, and local jurisdictions are investing hundreds of millions of dollars in retrofitting diesel engines in school buses and other changes to reach this goal.

The U.S. Environmental Protection Agency's recent regulations require all on-road diesel vehicles to change to low emission engines and ultra-low-sulfur fuels by 2007 (US EPA '00). In spring 2003, the U.S. EPA announced a nationwide voluntary school bus retrofit initiative. In July 2003, the Washington Legislature enacted a statewide "Diesel Solutions" program that provides 25 million dollars by 2008 to retrofit school diesel buses with cleaner burning engines and fuels, making it one of the largest and most active voluntary school bus retrofit program in the country. If risk assessment estimates are accurate, these changes will have a large public health impact, especially on children who ride school buses daily. However, no studies to-date have rigorously examined school children's exposure to diesel exhaust (DE) and its health effects, nor such a significant change in vehicular pollution control. We propose to seize this opportunity of a large natural experiment taking place in the Puget Sound area and conduct a study to assess health effects from diesel bus exhaust before and after the retrofit of diesel bus fleets between 2005 and 2007. The specific aims of the study are to:

1. Determine whether asthmatic children changing to retrofitted buses with cleaner fuels and engines have a reduction in sub-clinical and clinical asthma severity.
2. Determine if increased levels of DE exposure lead to an increase in acute clinical and sub-clinical features of asthma in children.
3. Quantify the levels and changes in particle and toxic gas exposures to DE in 3 groups of children commuting to school by retrofitted buses or private cars, old diesel buses to be retrofitted later, and old diesel buses through the study.

Sub-aim 3: Use the time-activity information, personal exposure measurements, and on-bus monitoring data to construct an exposure model to predict individual exposures to DE for all subjects.

DETAILED DESCRIPTION:
We will recruit 450 subjects ranging from 9 to 11 years old (or 3rd to 5th graders). These children who commute to school will perform repeated monthly measures of pulmonary function tests using spirometry, pulmonary inflammation via exhaled breath, and asthma symptoms and clinical encounters, up to 3 school years. These 500 children will represent 3 exposure scenarios: 1) one group of 125 children riding retrofitted school buses or private cars; 2) 250 children riding old buses who will change to retrofitted buses during the first or second year of the study; and 3) 125 children who ride old diesel buses through the study. All subjects will be either healthy or having physician-diagnosed asthma with severity ranging from mild intermittent to moderate persistent. Personal exposure monitoring of particulate matter, CO, NO2, and SO2 will be performed on a subset of 144 asthmatic subjects, with each subject being monitored for up to 2 days, in each monitoring year.

Subjects participating in the study will wear a small backpack containing several personal air monitors measuring real-time particulate matter concentrations and carbon monoxide concentrations as well as integrated (24 hour averaged) measurements of SO2 and NO2. The children's personal monitoring will begin when they wake up in the morning and continue for 24-hours. When wearing the backpack is inconvenient, such as when sleeping, the monitoring equipment should be placed in close proximity to the subject. Once the subject arrives at school, s/he will be asked to perform three respiratory tests: exhaled nitric oxide, exhaled breath condensate, and spirometry. At the end of the school day, the subject will be asked to perform the same two tests of lung function as earlier, plus an additional test of exhaled breath condensate. The subject will then continue his/her day as normal. A technician will replace the filter in the particulate matter monitor between 6 and 7 PM. We will repeat the same monitoring procedure the following morning when the subject wakes up for another 24-h. Monitoring will stop on the third morning when the subjects wake up. In addition to the personal monitoring, a monitoring kit will be installed in the subject's school bus and will be operated by a technician. This in-vehicle monitoring kit includes everything contained in the personal monitoring kit, plus a P-TRAK (TSI, model 8525) for real-time ultra-fine particle counts, two Harvard Personal Environmental Monitors (HPEM) with Teflon and quartz filters respectively for determining elemental carbon fractions, an EcoChem PAS2000CE monitor for polycyclic aromatic hydrocarbons (PAHs), and a global positioning system personal acquisition logger (GPS-PAL). The following timeline shows the typical daily schedule for a subject participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* ages 6-11 and attending 1st to 5th grades at schools in one of our target districts; approximately 75% subjects will commute by bus daily, 25% commute by car/walking;
* with or without physician-diagnosed asthma
* If with physician-diagnosed asthma:
* 1 year history, including episodic symptoms of wheezing, cough, and dyspnea;
* mild intermittent (with at least one episode a week requiring inhaler), mild persistent, or moderate persistent severity of asthma by NAEPP Criteria (NHLBI '91);

Exclusion Criteria:

* history of smoking by the subject or by a person in the subject's home
* asthma hospitalizations within 4 weeks of the start of each study year
* other chronic diseases such as diabetes, congenital heart disease, chronic renal disease
* new pets in the home

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2005-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L.-J. Sally Liu, Sc.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington Dept. Environmental and Occupational Health Sciences, Seattle, Washington, United States